CLINICAL TRIAL: NCT02643277
Title: A Pilot Study On The Effectiveness Of Using Automated Mobile Phone Text Messaging In Improving Glycaemic Control Among Newly Detected Type 2 Diabetic Patients
Brief Title: Effectiveness of Automated Mobile Phone Based Text Messaging on the Improvement of Glycaemic Outcomes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: India Diabetes Research Foundation & Dr. A. Ramachandran's Diabetes Hospitals (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IDRFARH001
Record Dates: First submitted 2015-01-16; First posted 2015-12-31 (Estimated); Last update posted 2019-04-02 (Actual); Status verified 2019-04

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Conventional care (Other): Conventional care is comprised of a one-to-one interview by a trained research personnel on diet and exercise advice at baseline and during every visit. The goals were to reduce portion size (total calories) and, to avoid simple sugars and refined carbohydrates, reduce total fat intake, restrict use of saturated fat, include more fibre rich food-(e.g., whole grains, legumes, vegetables, and fruits).
  Interventions: Other: Conventional care
- Mobile phone text messaging (Experimental): The intervention will receive text messages delivered by an automated text messaging manager. The message content will be designed to induce lifestyle modification (diet and physical activity) and will be motivational, based on the content which has been proven to be effective in reducing progression to diabetes in people with pre-diabetes. Other text messages will aim to improve drug compliance and disease monitoring. The messages provide tips and suggestions, and positive reinforcement or encouragement, for improving lifestyle behaviors and compliance with therapy.
  Interventions: Behavioral: Mobile phone text messaging

INTERVENTIONS:
Behavioral: Mobile phone text messaging — The intervention will be text messages delivered by an automated text messaging manager. The message content will be designed to induce lifestyle modification (diet and physical activity) and will be motivational, based on the content which has been proven to be effective in reducing progression to diabetes in people with pre-diabetes. Other text messages will aim to improve drug compliance and disease monitoring, based on our pilot studies in India. The control arm will receive conventional management, according to local guidelines in the Indian centers, which in all cases are compatible with those of the International Diabetes Federation.
  Arms: Mobile phone text messaging
Other: Conventional care — Conventional care is comprised of a one-to-one interview by a trained research personnel on diet and exercise advice at baseline and during every visit. The goals were to reduce portion size (total calories) and, to avoid simple sugars and refined carbohydrates, reduce total fat intake, restrict use of saturated fat, include more fibre rich food-(e.g., whole grains, legumes, vegetables, and fruits).
  Arms: Conventional care

SUMMARY:
In India, the high diabetes prevalence and cost of its management relative to their personal income render the country an appropriate environment to seek and test new, less expensive aids to care. Education and motivation to induce behavioural modification, are important components of care. Conventional diabetes education programmes involving personal contact methods are useful but expensive. Compliance with medications is also important and there are data to suggest that compliance is low in people with established type 2 diabetes (there is little information on those with recently diagnosed disease). Mobile phones could provide an inexpensive and scaleable delivery vehicle for components of care. There are now more than 5 billion wireless subscribers and 70% of them live in low and middle income countries. Mobile phone ownership is high in India and an increasing proportion now has Mobile phones and/or home computers. The investigators plan a clinical trial in India to assess whether there is benefit from an enhanced text message intervention delivered by mobile phone in people newly diagnosed with Type 2 diabetes. The message content will be directed to behavioural modification, as with our diabetes prevention studies, and will attempt to improve compliance with drug therapy and other aspects of care, as with our studies in people with established diabetes. The investigators shall compare effects on glycaemia, other cardiovascular risk factors, lifestyle behaviour and quality of life, with those observed in people with type 2 diabetes receiving standard care.

DETAILED DESCRIPTION:
India currently has 65 million people with type 2 diabetes and the number is increasing. In addition to its human costs, diabetes imposes a large economic burden. In those of average income in India, diabetes care consumes 25% of the family budget where one member is affected and proportionately more when there are other affected members (which is not uncommon); much of this expenditure is on medical and nursing costs aimed at achieving good glycaemic control. Diabetes management is important because it leads to better long-term clinical outcomes. The proof of principle trial - United Kingdom Prospective Diabetes Study (UKPDS) in patients with type 2 diabetes demonstrated that glycaemic control from the time of diagnosis produced beneficial effects during the trial and that these persisted for at least ten years afterwards (despite the confluence of HbA1c levels post-trial). There was continued improvement in microvascular complications and emergent significant reductions in myocardial infarction and death - the 'legacy effect'. Similar prolonged benefit has been demonstrated for Type 1 diabetes in the Diabetes Control and Complication Trial (DCCT) and its follow-up (for at least 17 years).

Improving glycaemic control involves lifestyle modification (diet and physical activity), prompt introduction of hypoglycaemic therapy where necessary and then compliance with the treatment and monitoring. Dietary measures early after diagnosis lead to improved glycaemia and reductions in other cardiovascular risk factors. The importance of physical activity is often overlooked, but it contributes to maintenance of weight loss long-term, improves physical fitness and reduces cardiovascular risk factors. At or shortly after diagnosis, diabetes education aiming at lifestyle change is helpful in modifying behaviour and can reduce HbA1c. Although these programmes are effective, the benefits diminished over time e.g. the DESMOND programme resulted in improved HbA1c levels at twelve months but not at three years. There is evidence that the sustained benefit may be more likely if the educational programme is reinforced at a later stage. A major barrier to implementation of all education programmes, and particularly those which include reinforcement, is cost. Because they involve personal contact, the programmes are expensive and in reality, are offered to only small proportion of patients, even in developed countries. Although attempts have been made to utilise trained non-medical, non-nursing staff in education programmes in India, this model, while less expensive, has not been widely adopted. Attendance at educational sessions is also problematic, as it requires taking time off work or away from the family, or the venue is considered inaccessible.

Text messaging (short message service, SMS) has the potential to overcome some of the difficulties. It is relatively cheap and potentially scalable. For example, in people with pre-diabetes in India the investigators have shown a 36% reduction in progression to diabetes over 2 years with text messaging-assisted behavioural modification. This reduction is similar to that achieved in India using personal contact methods. There are relatively few high quality studies on the role of text messaging or mobile phone contact as an aid to management of established Type 2 diabetes. In a pilot study in India, the investigators have demonstrated that text messaging can improve compliance with medications. A recent Cochrane review of IT-assisted methodologies for diabetes care and education suggested a small benefit for glycaemia, greatest where mobile phones (as opposed to home computers) were the delivery medium. The average lowering of HbA1c, as a result of mobile phone input on a range of studies was 5.5 mmol/mol (0.5%). This is clinically significant. Part of the reason for this benefit may reside in the nature of mobile phone contacts, being passive and, if appropriately designed, the message content can be encouraging rather than threatening in nature. The messages can also be sent repeatedly, with their frequency and timing dictated by the recipient.

ELIGIBILITY:
Inclusion Criteria:

1. Newly diagnosed Type 2 Diabetes Mellitus patients not receiving any medication for diabetes.
2. Patients who consent to participate in the study
3. Both sexes of age ≥ 20 and ≤ 60 years.
4. Having an HbA1c level of ≥ 6.5 % (48 mmol/mol) on diagnosis
5. Willing to report periodically for investigations during the study period
6. Ability to read and understand messages.

   -

Exclusion Criteria:

1. Type 1 Diabetes
2. Major illness - such as Cancer, Cardiovascular Disease, Chronic liver or kidney disease on diagnosis of diabetes.
3. Disorders with cognitive impairment, severe depression or mental imbalance.
4. Physical disability that would prevent regular physical activity.
5. Participants unwilling to participate in the study.
6. Participants who do not possess a mobile phone.
7. Participants not able to read and understand SMS.
8. Participants below the age of 20 years and above the age of 60 years.

   -

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 244 (Actual)
Dates: Start 2014-12 (Actual); Primary Completion 2018-04 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Comparison of the glycaemic outcome measured as improvement in HbA1c (≤ 7.0% (53mmol/mol)) in the intervention group in comparison with the conventional care. | 2 years

SECONDARY OUTCOMES:
Changes in body mass index | Baseline and 2 years
  We are assessing the changes in BMI not the changes in weight & height and the unit for BMI is Kg/m2. It is a single unit of measurement calculated by patients weight and Height.
Changes in blood pressure | Baseline and 2 years
Changes in fasting and postprandial plasma glucose | Baseline and 2 years
Changes in lipid profile | Baseline and 2 years
Improvement in quality of life | Baseline and 2 years
  Scale
Improvement in acceptance of this strategy as an educative tool by the patients | Baseline and 2 years
  Questionnaire
Adherence to the prescription | Baseline and 2 years
  Analysis

CONTACTS AND LOCATIONS:
Overall Officials: Ambady Ramachandran, Prof, Principal Investigator — Chairman, India Diabetes Research Foundation
Locations (1):
- Dr.A.Ramachandran's Diabetes Hospitals, Chennai, Tamil Nadu, India

IPD SHARING:
Plan to Share IPD: Undecided